CLINICAL TRIAL: NCT07158229
Title: Social and Psychological Long-term Impact of NMDA Receptor Encephalitis, Level 3
Brief Title: Long-term Impact of NMDAR Encephalitis, Level 3
Acronym: SAPIENCE 3
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0541
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: NMDAR Autoimmune Encephalitis
Keywords: NMDAR encephalitis; psychosocial impact
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-NMDAR encephalitis patients: Patients over 18 years old with NMDAR encephalitis.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Complete quality of life questionnaires focusing on fatigue, anxiety, depression, and sleep.

SUMMARY:
NMDA receptor antibody encephalitis is a rare autoimmune neurological disease of the central nervous system with an estimated incidence of 1.5 people per million per year. Patients with anti-NMDAR encephalitis experience an acute phase of the disease characterized by psychosis, memory loss, seizures, autonomic nervous system instability, or coma. Since the discovery of this disease 14 years ago by Prof. Dalmau, the clinical presentation of the acute phase has been well characterized, while the psychosocial impact of the disease remains largely unexplored.

Currently, there are few cohort studies of patients that have identified persistent cognitive impairment as a factor impacting remission after the acute phase. Given the scarcity of information concerning the post-acute phase, it is therefore essential to determine the long-term social and psychological outcomes and their daily effects on the social and functional life of this severe disease. This is especially important as the patients are young, with a median age of 21 years, and may face lasting limitations potentially detrimental to their success in professional, educational, or social environments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NMDAR encephalitis
* Age ≥ 18 years old
* Patient affiliated to a social security system
* No opposition from the patient
* Access to an internet connection and a computer

Exclusion Criteria:

* Patients whithout NMDAR encephalitis
* Patient under guardianship or curatorship
* Patient with neurological disorders pre-existing encephalitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anti-NMDA encephalitis aged over 18 years old and followed throughout France.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of cognitive assessments and psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease - PREMS questionnaires - AEPREM questionnaire | At inclusion
  AEPREM questionnaire (stands for "evaluation of experience in healthcare facilities and medical teams" in french)
Analysis of cognitive assessments and psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease - PREMS questionnaire - AESOC | At inclusion
  AESOC questionnaire ( stands for "questionnaire on clinical symptoms and perception of the disease" in french)
Analysis of cognitive assessments and psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease - PROMS questionnaires - FSS questionnaire | At inclusion
  FSS questionnaire (stands for "fatigue severity scale") assesses fatigue in patients. Questionnaire is composed of 9 items graded on a scale from 1 to 7. Score varies from 9 to 63. The higher the score, the strongest the fatigue.
Analysis of cognitive assessments and psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease - PROMS questionnaire - GAD7 | At inclusion
  GAD7 questionnaire (stands for "Generalized Anxiety Disorder 7") assesses anxiety in patients. Items are rated on a scale of 0 to 3. Score varies from 0 to 21. The recommended threshold for estimating generalised anxiety is 10.
  Thresholds:
  No anxiety: 0-4 points; Mild anxiety: 5-9 points; Moderate anxiety: 10-14 points; Severe anxiety: 15-21 points.
Analysis of cognitive assessments and psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease - PROMS questionnaire - PHQ9 questionnaire | At inclusion
  PHQ9 questionnaire (stands for "Patient Health Questionnaire-9") assesses depression in patients. Questionnaire is composed of 9 items each graded from 0 to 3. Score varies from 0 to 27. The higher the score, the more depressed is the patient.
Analysis of cognitive assessments and psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease - PROMS questionnaire - PSQI questionnaire | At inclusion
  PSQI questionnaire (stands for "Pittsburgh Sleep Quality Index") assesses sleep in patients. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
Analysis of cognitive assessments and psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease - PROMS questionnaire - EQ-5D-5L questionnaire | At inclusion
  EQ-5D-5L questionnaire (stands for "EuroQol-5-Dimension") assesses quality of life in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologies paranéoplasiques et encéphalites auto-immunes - Hôpital neurologiques Pierre WERTHEIMER - Groupement hospitalier Est - Hospices civiles de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No